CLINICAL TRIAL: NCT00800865
Title: A 2-Stage, Open Label, Phase Ib Clinical Trial to Evaluate Biomarkers in Patients With Solid Tumor and Receiving a Single Dose of Cytotoxics
Brief Title: A Study to Evaluate Biomarkers in Patients With Solid Tumors (0000-097)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-097; 2008_593
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biomarker Evaluation Group I (Other): Biomarker evaluation before and after dosing with cytotoxic agent(s)
  Interventions: Other: Biomarker sample collection before and after dosing with cytotoxic agent(s)
- Biomarker Evaluation Group II (Other): Biomarker evaluation before and after dosing with cytotoxic agent(s)
  Interventions: Other: Biomarker sample collection before and after dosing with cytotoxic agent(s)

INTERVENTIONS:
Other: Biomarker sample collection before and after dosing with cytotoxic agent(s) — Participants will have blood and urine samples collected at Visit 1. After allocation, punch skin biopsies, plucked hair samples, blood, and urine will be collected at baseline, and at 24 and 48 hours post dosing with cytotoxic agent(s).
  Arms: Biomarker Evaluation Group I
Other: Biomarker sample collection before and after dosing with cytotoxic agent(s) — A second group of participants will have blood and urine samples collected at Visit 1 (there is no baseline). After allocation, punch skin biopsies, plucked hair samples, blood, and urine will be collected at at 24, 32 and 48 hours post dosing with cytotoxic agent(s).
  Arms: Biomarker Evaluation Group II

SUMMARY:
A study to evaluate biomarkers of cancer (context-specific sensitizers) in the skin of participants already receiving cytotoxic therapy. Additional blood and urine samples will be collected for phosphorylated Histone 2AX (γH2AX) and renal toxicity biomarker testing, respectively.

ELIGIBILITY:
Inclusion Criteria:

Participant has solid tumor that will be treated with one of the following treatments:

* Gemcitabine monotherapy
* Cisplatin monotherapy
* Carboplatin monotherapy
* Gemcitabine and cisplatin combination therapy
* Gemcitabine and erlotinib combination therapy
* Gemcitabine and carboplatin combination therapy
* Cisplatin and vinorelbine combination therapy
* Cisplatin and pemetrexed combination therapy
* Carboplatin and vinorelbine combination therapy
* Carboplatin and pemetrexed combination therapy

Exclusion Criteria:

* Participant has had recent cancer treatments including chemotherapy or radiation
* Participant has been in an investigational study within the last 30 days
* Participant has a history of drug or alcohol abuse
* Participant is Human Immunodeficiency Virus (HIV) positive or has a history of Hepatitis B or C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Sun A, Lam R, Harman A, Pavlick A, Herman G, Dauffenbach L, Kerfoot C, Huang P, Cheng J, Demuth T, Iannone R. Induction of CDC2 phosphylation in skin biopsies from patients with solid tumors undergoing DNA-damaging chemotherapy. Global J Med Res. 2014;14(1-K):11-21

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 36 participants enrolled. Of these, 4 from Group I and 1 from Group II did not have evaluable biopsies and were considered not evaluable. Data only reflect the evaluable population (15 from Group I and 16 from Group II).
Groups:
- Biomarker Evaluation Group I: Participants who had blood and urine samples collected at Visit 1. After allocation, punch skin biopsies, plucked hair samples, blood, and urine were collected at baseline, and at 24 and 48 hours post dosing with cytotoxic agent(s). An additional sample collection at 32 hours may have been performed if deemed necessary after review of the data.
- Biomarker Evaluation Group II: A second group of participants who had blood and urine samples collected at Visit 1 (there was no baseline). After allocation, punch skin biopsies, plucked hair samples, blood, and urine were collected at at 24, 32 and 48 hours post dosing with cytotoxic agent(s).
Period: Overall Study
Arm/Group | Biomarker Evaluation Group I | Biomarker Evaluation Group II
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biomarker Evaluation Group I | Biomarker Evaluation Group II | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Customized [Number; unit: participants]
  29-77 years | 15 | 0 | 15
  34-88 years | 0 | 16 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Level of Biomarkers
Description: Phospho-CDC2 (pCDC2) response in the skin following the administration of cytotoxic agents. pCDC2 levels were measured by immunohistochemistry (IHC).
Time Frame: Baseline, 24, 32, and 48 hours post dose
Population: Actual number of participants analyzed in Part I varied from 13 to 15, depending on time point. Actual number of participants analyzed in Part II was 16 for all time points.
Measure: Geometric Mean (90% Confidence Interval); unit: Percent pCDC2-positive cells
Arm/Group | Biomarker Evaluation Group I | Biomarker Evaluation Group II
Number analyzed (Participants) | 15 | 16
Percent pCDC2-positive cells
  Baseline | 24.6 (1.7) [19.0 to 31.8] | NA (NA) [NA to NA] — Baseline value is not applicable in Part II
  24 hours post chemotherapy | 34.3 (1.9) [25.6 to 46.0] | 23.0 (1.9) [17.4 to 30.3]
  32 hours post chemotherapy | NA (NA) [NA to NA] — No samples taken at this time point in Part I | 23.7 (2.0) [17.5 to 32.1]
  48 hours post chemotherapy | 50.3 (1.7) [39.9 to 63.5] | 29.9 (1.8) [23.2 to 38.6]

2. Primary Outcome: Ratio of pCDC2 Response in Skin Following Administration of Cytotoxic Therapy
Description: Ratio of Phospho-CDC2 (pCDC2) response at 24, 32, and 48 hours compared to baseline, 24, and 32 hours post chemotherapy.
Time Frame: 24, 32, and 48 hours post dose
Measure: Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Biomarker Evaluation Group I | Biomarker Evaluation Group II
Number analyzed (Participants) | 15 | 16
Ratio
  24 hours post chemotherapy/baseline | 1.40 (1.59) [1.11 to 1.75] | NA (NA) [NA to NA] — Ratio not applicable for Part II
  48 hours post chemotherapy/baseline | 2.05 (1.78) [1.56 to 2.69] | NA (NA) [NA to NA] — Ratio not applicable for Part II
  32 hours/24 hours post chemotherapy | NA (NA) [NA to NA] — Ratio not applicable for Part I | 1.03 (1.60) [0.84 to 1.27]
  48 hours/24 hours post chemotherapy | 1.47 (NA) [1.12 to 1.91] | 1.30 (1.80) [1.01 to 1.69]
  48 hours/32 hours post chemotherapy | NA (NA) [NA to NA] — Ratio not applicable for Part I | 1.26 (1.75) [0.99 to 1.62]

ADVERSE EVENTS:
Arm/Group | Biomarker Evaluation Group I | Biomarker Evaluation Group II
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 4/15 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biomarker Evaluation Group I (N=15) | Biomarker Evaluation Group II (N=16)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This is an exploratory study to develop data for possible future studies. It is not intended to be published, unless important new information or data concerning the safety of a marketed product is obtained. The Sponsor must have the opportunity to review all abstracts, manuscripts, or presentations 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. Sponsor review can be expedited.